CLINICAL TRIAL: NCT01621646
Title: The Effect of Consumption of 2 Eggs or 4 oz of Egg Substitute Daily for 6 Months on Cognitive Function in Older Adults.
Brief Title: The Effect of Daily Consumption of Eggs on Cognitive Function in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2012-03-13; First posted 2012-06-18 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Mild Cognitive Impairment
Keywords: lutein; eggs; mild cognitive impairment; elderly
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Eggs; Egg White

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- egg white (control) (Placebo Comparator): egg whites, 4 ounces per day for six months
  Interventions: Other: eggs or egg whites
- eggs (Experimental): eggs, 2 large per day for 6 months
  Interventions: Other: eggs or egg whites

INTERVENTIONS:
Other: eggs or egg whites — 2 eggs/day or 4 oz egg whites/day for 6 months

SUMMARY:
Cognitive impairment is also a major risk factor for development of dementia later in life. Findings from our studies suggest that the carotenoids, lutein and zeaxanthin may be important in cognitive function in the elderly. The investigators have previously reported eggs to be a highly bioavailable source of lutein and zeaxanthin. Our study evaluates long-term egg intervention as a treatment strategy for age-related cognitive impairment which could possibly prevent the onset of dementia. The investigators have also shown that lutein supplementation significantly improved verbal fluency scores in healthy older women. Our studies have shown that egg interventions can significantly increase serum lutein concentrations in older adults. Based on the sum of our findings, the next logical step will be to investigate the ability of lutein and zeaxanthin contained in eggs to influence cognitive function in older adults. The investigators hypothesize that there will be a significant increase in cognitive function measures in older adults provided with meals containing 2 egg/day at the end of 6 months, while no significant improvements will be observed in older adults given daily meals containing egg substitute.

The proposed study is designed as a randomized, placebo controlled trial that tests the effects of 6 month supplementation with 2 eggs/day on cognitive function in older adults. Secondary analyses will determine whether baseline MP density predicts relative effectiveness of the intervention on cognitive function. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation.

DETAILED DESCRIPTION:
The study is designed as a placebo controlled trial that tests the effects of 6 month supplementation with 2 eggs or 4 ounces of egg substitute a day on cognitive function in older adults. Subjects will be randomly assigned to one of the two groups. Secondary analyses will determine whether baseline macular pigment density (a non invasive measure of lutein and zeaxanthin in neural tissue) or choline status predicts relative effectiveness of the intervention on cognitive function. Secondary outcomes include plasma biomarkers of oxidative stress and inflammation, choline bioavailability, and genetic variants related to endogenous choline production. Participants will be recruited from community-dwelling men and women aged > 50 yr, and potential participants will be screened to meet cognitive and functional criteria. Participants will be pre-screened by telephone; those who appear to meet criteria will undergo further screening. The study will include baseline (0 month), 3 and 6 month visits for study procedures, and monthly telephone calls. Given that there is a visible difference between the two interventions (eggs, egg substitute), a blinded study is not possible.

ELIGIBILITY:
Inclusion Criteria:

* men and women age > 50 years
* BMI 19-30 kg/m2
* lutein intake of < 3 mg/d
* DHA (docosahexaehoic acid) intake < 250 mg/d (including supplements)
* Mini mental state exam (MMSE) score > 24 (Appendix B)
* macular pigment density < 0.5 at 0.5 degrees
* Beck Depression Inventory < 20
* free of known disease;
* BMI 19-29 kg/m2
* must be able to give written informed consent
* have normal hematologic parameters
* normal values of plasma albumin
* normal values for liver and kidney function (Appendix A)
* no use of carotenoid, n3 fatty acid, multivitamin/mineral, or choline supplements (> 3 months).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
cognition | 6 months
  measures of attention, executive function, verbal fluency will be made using a sensitive computerized program

SECONDARY OUTCOMES:
inflammation | 6 months
  markers of inflammation will be made in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Johnson, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States